CLINICAL TRIAL: NCT04369300
Title: Prevalence Of Anxiety And Depression During COVID-19
Brief Title: Anxiety And Depression During COVID-19 IN INDIA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Max Healthcare Insititute Limited (Other)
Responsible Party: Sponsor
Other Study IDs: Covid-19/MHC/PSYCH/20-10
Record Dates: First submitted 2020-04-28; First posted 2020-04-30 (Actual); Last update posted 2020-07-15 (Actual); Status verified 2020-07

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Registery Data Collection — Observational Data Collection

SUMMARY:
1. To understand the prevalence of symptoms of Depression and Anxiety in general population during COVID-19 in India
2. To understand correlation between COVID-19 related factors and mental health symptomology in the general population in India

Hypothesis:

There is likelihood of significant symptoms of depression and anxiety among general population in India during the current COVID-19 outbreak.

Procedure:

The participants would be selected with their informed consent. The objective of the study would be clearly written on Page 1 of the survey. The test would be administered electronically by all the participants individually only when consented to the study. The data collected will be kept strictly confidential and the identity of the participants will not be disclosed at any point of the research

Measures:

1. Demographic Information Demographic variables included Gender, Age, Place of Stay, Marital Status, Highest Level ofEducation, current living arrangement (e.g. staying alone or with family) and Occupation. It further includesregular employment status and current employment status(e.g, Work from home, temporary leave, termination etc)
2. History of illness (Present or past) History of physical ailment specified (diabetes, hypertension, heart ailment or being on any steroid or any other chronic ailment) Previous history of H1N1/ Influenza like illness
3. COVID-19 Information This section includes time spent focusing on COVID related information, current stressors with respect to COVID-19 and coping mechanisms used. This further includesinformation on resources available to participants near their place of stay and information of any known diagnosed case of COVID-19.
4. Standardized Scales to be used Generalized Anxiety Disorder Scale (GAD-7); Patient Health Questionnaire (PHQ-9) Powered by

DETAILED DESCRIPTION:
Aim:

1. To understand the prevalence of symptoms of Depression and Anxiety in general population during COVID-19 in India
2. To understand correlation between COVID-19 related factors and mental health symptomology in the general population in India

Hypothesis:

There is likelihood of significant symptoms of depression and anxiety among general population in India during the current COVID-19 outbreak.

Procedure:

The participants would be selected with their informed consent. The objective of the study would be clearly written on Page 1 of the survey. The test would be administered electronically by all the participants individually only when consented to the study. The data collected will be kept strictly confidential and the identity of the participants will not be disclosed at any point of the research

Measures:

1. Demographic Information Demographic variables included Gender, Age, Place of Stay, Marital Status, Highest Level of Education, current living arrangement (e.g. staying alone or with family) and Occupation. It further includes regular employment status and current employment status(e.g, Work from home, temporary leave, termination etc)
2. History of illness (Present or past) History of physical ailment specified (diabetes, hypertension, heart ailment or being on any steroid or any other chronic ailment) Previous history of H1N1/ Influenza like illness
3. COVID-19 Information This section includes time spent focusing on COVID related information, current stressors with respect to COVID-19 and coping mechanisms used. This further includes information on resources available to participants near their place of stay and information of any known diagnosed case of COVID-19.
4. Standardized Scales to be used Generalized Anxiety Disorder Scale (GAD-7); Patient Health Questionnaire (PHQ-9)

Primary outcome To understand the prevalence (magnitude) of depression and anxiety of general adult population during COVID-19 using Generalized Anxiety Disorder Scale (GAD-7) and Patient Health Questionnaire (PHQ-9). Rise in Anxiety and Depression will be noted.

Through the analysis of the results, help device psychological intervention/mental health programs geared towards general and specific symptoms and management of emotional needs can be provided to the general population during and post-crisis.

Secondary Outcome Through the analysis of the results, it will help device psychological intervention/mental health programs geared towards general and specific symptoms and management of emotional needs can be provided to the general population during and post-crisis.

ELIGIBILITY:
Inclusion Criteria:

* Participants of the age of 18 years and above
* Participants residing in India
* Participants with minimum 10 years of education with basic knowledge of English

Exclusion Criteria:

* Participants under the age of 18 years
* Participants residing outside of India
* Participants with previous history of any major psychiatric illness, psychiatric hospitalization or currently on any psychiatric medication.

Ages: 18 Years to 90 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Participants of the age of 18 years and above
  Participants residing in India
  Participants with minimum 10 years of education with basic knowledge of English
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2020-04-24 (Actual); Primary Completion 2020-11-24 (Estimated); Study Completion 2021-02-24 (Estimated)

PRIMARY OUTCOMES:
Prevalence (magnitude) of anxiety of general adult population during COVID-19 | 1 YEAR
  To understand the prevalence (magnitude) of depression and anxiety of general adult population during COVID-19 using Generalized Anxiety Disorder Scale (GAD-7)
prevalence (magnitude) of depression and anxiety of general adult population during COVID 19 | 1 Year
  To understand the prevalence (magnitude) of depression and anxiety of general adult population during COVID-19 using Patient Health Questionnaire (PHQ-9).

CONTACTS AND LOCATIONS:
Overall Officials: Sameer Malhotra, Principal Investigator — max healthcare
Locations (1):
- Max Super Speciality hospital, New Delhi, National Capital Territory of Delhi, India